CLINICAL TRIAL: NCT00686543
Title: A Phase 4 Study of the Pharmacokinetics of Oral Posaconazole (SCH 56592) Among Patients With Compromised Gastrointestinal Function and at High Risk for Invasive Fungal Infection
Brief Title: Oral Posaconazole in High Risk Patients With Gastrointestinal Dysfunction (Study P05115)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P05115; EudraCT No. 2007-003148-31
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Fungal Infection; Acute Myelogenous Leukemia; Neutropenia
Keywords: Antifungal Agents; Anti-Infective Agents
MeSH Terms: conditions — Mycoses; Leukemia, Myeloid, Acute; Neutropenia | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- POS 200 mg TID Days 1-8 Followed by POS 200 mg TID Days 9-15 (Experimental): POS 200 mg three times a day (TID) on Days 1-8 followed by continued randomized dosing regimen of POS 200 mg TID on Days 9-15, administered with food or oral nutritional supplements.
  Interventions: Drug: Posaconazole
- POS 200 mg TID Days 1-8 Followed by POS 400 mg BID Days 9-15 (Experimental): POS 200 mg TID on Days 1-8 followed by randomized dosing regimen of POS 400 mg twice a day (BID) on Days 9-15, administered with food or oral nutritional supplements.
  Interventions: Drug: Posaconazole
- POS 200 mg TID Days 1-8 Followed by POS 400 mg TID Days 9-15 (Experimental): POS 200 mg TID on Days 1-8 followed by randomized dosing regimen of POS 400 mg TID on Days 9-15, administered with food or oral nutritional supplements.
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — Posaconazole will be used for prophylaxis
  Other Names: SCH 056592 - NOXAFIL®

SUMMARY:
The purpose of this study is: to explore the potential for different dosing strategies of posaconazole oral suspension (POS) to increase plasma levels and to profile the pharmacokinetics of these dosing strategies in patients with compromised gastrointestinal function and at high risk for Invasive Fungal Infection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >=18 years of age
* High risk of poor enteral medication absorption, based on the effects of cytotoxic chemotherapy, as evidenced by, but not limited to, mucositis, nausea, vomiting, and diarrhea, at baseline.
* High risk of invasive fungal infection (IFI) based on anticipated or documented prolonged neutropenia (absolute neutrophil count [ANC] <500/mm^3 [0.5 x 10^9/L]).
* Clinical laboratory safety tests within normal limits or clinically acceptable to the investigator or sponsor.
* Free of any clinically significant disease (other than the primary hematologic disease) that would interfere with the study evaluations.
* Subjects must be willing to give written informed consent and able to adhere to dosing, study visit schedule, and mandatory procedures.

Exclusion Criteria:

* Female subjects who are pregnant, intend to become pregnant, or are nursing.
* Excluded prior treatments. Subjects receiving systemic antifungal therapy (oral, intravenous, or inhaled) for the treatment of proven or probable IFI within 30 days of Enrollment (ie, voriconazole, fluconazole [FLU], or itraconazole [ITZ]).
* Subjects receiving posaconazole for prophylaxis against IFI 10 days prior to enrollment. (Subjects who are receiving either voriconazole or micafungin for prophylaxis against IFI should discontinue those therapies upon enrollment.)
* Subjects with moderate or severe liver dysfunction at Baseline, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels greater than two times the upper limit of normal (ULN), or a total bilirubin level greater than two times the ULN.
* Subjects who have taken prohibited medications more recently than the indicated washout period prior to Enrollment.
* Subjects who must take prohibited medications during the study.
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Subjects who have used any investigational drugs or biologic agents other than their chemotherapy regimens within 30 days of study entry.
* Subjects who are part of the staff personnel directly involved with this study.
* Subjects who are a family member of the investigational study staff.
* Prior enrollment in this study.
* Subjects with a history of hypersensitivity or idiosyncratic reactions to azole agents.
* Subjects with Eastern Cooperative Oncology Group (ECOG) performance status >2 prior to induction chemotherapy for their underlying disease.
* Subjects with proven or probable invasive or systemic fungal infection at Baseline.
* Subjects with a history of acute lymphoblastic leukemia or chronic myelogenous leukemia without blast crisis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Cornely OA, Helfgott D, Langston A, Heinz W, Vehreschild JJ, Vehreschild MJ, Krishna G, Ma L, Huyck S, McCarthy MC. Pharmacokinetics of different dosing strategies of oral posaconazole in patients with compromised gastrointestinal function and who are at high risk for invasive fungal infection. Antimicrob Agents Chemother. 2012 May;56(5):2652-8. doi: 10.1128/AAC.05937-11. Epub 2012 Jan 30. PMID 22290953

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Randomized: Posaconazole oral suspension (POS) 200 mg Three Times a Day (TID) on Days 1-8, administered with food or oral nutritional supplements (participants who discontinued anytime before randomization on Day 8)
- POS 200 mg TID Days 1-8 Followed by POS 200 mg TID Days 9-15: POS 200 mg TID on Days 1-8 Followed by POS 200 mg TID on Days 9-15, administered with food or oral nutritional supplements (participants who received POS 200 mg TID on Days 1-8 and were then randomized to continue with POS 200 mg TID on Days 9-15).
- POS 200 mg TID Days 1-8 Followed by POS 400 mg BID Days 9-15: POS 200 mg TID on Days 1-8 followed by POS 400 mg Twice a Day (BID) on Days 9-15, administered with food or oral nutritional supplements (participants who received POS 200 mg TID on Days 1-8 and were then randomized to POS 400 mg BID on Days 9-15).
- POS 200 mg TID Days 1-8 Followed by POS 400 mg TID Days 9-15: POS 200 mg TID on Days 1-8 followed by POS 400 mg TID on Days 9-15, administered with food or oral nutritional supplements (participants who received POS 200 mg TID on Days 1-8 and were then randomized to POS 400 mg TID on Days 9-15).
Period: Overall Study
Arm/Group | Not Randomized | POS 200 mg TID Days 1-8 Followed by POS 200 mg TID Days 9-15 | POS 200 mg TID Days 1-8 Followed by POS 400 mg BID Days 9-15 | POS 200 mg TID Days 1-8 Followed by POS 400 mg TID Days 9-15
Started | 14 | 21 | 20 | 20
Completed | 0 | 20 | 15 | 17
Not Completed | 14 | 1 | 5 | 3
Not completed — Adverse Event | 9 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: POS 200 mg TID on Days 1-8, administered with food or oral nutritional supplements (participants who discontinued anytime before randomization on Day 8).
- POS 200 mg TID Days 1-8 Followed by POS 400 mg BID Days 9-15: POS 200 mg TID on Days 1-8 followed by POS 400 mg BID on Days 9-15, administered with food or oral nutritional supplements (participants who received POS 200 mg TID on Days 1-8 and were then randomized to POS 400 mg BID on Days 9-15).
- Total: Total of all reporting groups
Arm/Group | Not Randomized | POS 200 mg TID Days 1-8 Followed by POS 200 mg TID Days 9-15 | POS 200 mg TID Days 1-8 Followed by POS 400 mg BID Days 9-15 | POS 200 mg TID Days 1-8 Followed by POS 400 mg TID Days 9-15 | Total
Number analyzed (Participants) | 14 | 21 | 20 | 20 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 16 | 16 | 19 | 62
  >=65 years | 3 | 5 | 4 | 1 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 11 | 9 | 36
  Male | 8 | 11 | 9 | 11 | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean POS Plasma Concentrations on Days 2, 3, and 8.
Description: Individual mean concentrations were calculated as the average of observed concentrations at 0 hour (before the morning dose) and 5 hours after the morning dose.
Time Frame: Predose (0 hour) and 5 hours postdose on Days 2, 3, and 8
Population: Analysis of the primary outcome was done on the Balanced Data Set, defined as all participants with no missing pharmacokinetic data for Days 3, 8, and 15 (n=49). From Days 1 to 8, these 49 participants received 200 mg TID. From Days 9 to 15, these 49 participants were randomized to either 200 mg TID (n=19), 400 mg BID (n=14), or 400 mg TID (n=16).
Measure: Mean (90% Confidence Interval); unit: ng/mL
Groups:
- POS 200 mg TID Days 1-8: POS 200 mg TID on Days 1-8, administered with food or oral nutritional supplements (participants who received POS 200 mg TID on Days 1-8 and were then randomized to one of the three dosing regimens for Days 9-15).
Arm/Group | POS 200 mg TID Days 1-8
Number analyzed (Participants) | 49
ng/mL
  Day 2 | 230 [194 to 266]
  Day 3 | 346 [296 to 396]
  Day 8 | 637 [521 to 753]

2. Primary Outcome: Mean POS Plasma Concentrations on Days 8 and 15 Stratified by Randomized Dosing Regimen
Description: as for outcome 1
Time Frame: Predose (0 hour) and 5 hours postdose on Days 8 and 15
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | POS 200 mg TID Days 1-8 Followed by POS 200 mg TID Days 9-15 | POS 200 mg TID Days 1-8 Followed by POS 400 mg BID Days 9-15 | POS 200 mg TID Days 1-8 Followed by POS 400 mg TID Days 9-15
Number analyzed (Participants) | 19 | 14 | 16
ng/mL
  Day 8 | 620 [439 to 800] | 849 [541 to 1156] | 473 [361 to 585]
  Day 15 | 660 [487 to 834] | 930 [617 to 1243] | 671 [530 to 811]

3. Primary Outcome: Participants With a Mean POS Plasma Concentration ≥/<250 ng/mL on Day 3 and ≥/<500 ng/mL on Day 8
Description: as for outcome 1
Time Frame: Predose (0 hour) and 5 hours postdose on Days 3 and 8
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | POS 200 mg TID Days 1-8
Number analyzed (Participants) | 49
Participants
  Day 3 <250 ng/mL and Day 8 <500 ng/mL | 17
  Day 3 <250 ng/mL and Day 8 ≥500 ng/mL | 2
  Total Day 3 <250 ng/mL | 19
  Day 3 ≥250 ng/mL and Day 8 <500 ng/mL | 8
  Day 3 ≥250 ng/mL and Day 8 ≥500 ng/mL | 22
  Total Day 3 ≥250 ng/mL | 30

4. Primary Outcome: Participants With a Mean POS Plasma Concentration ≥/<350 ng/mL on Day 3 and ≥/<700 ng/mL on Day 8
Description: as for outcome 1
Time Frame: Predose (0 hour) and 5 hours postdose on Days 3 and 8
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | POS 200 mg TID Days 1-8
Number analyzed (Participants) | 49
Participants
  Day 3 <350 ng/mL and Day 8 <700 ng/mL | 25
  Day 3 <350 ng/mL and Day 8 ≥700 ng/mL | 3
  Total Day 3 <350 ng/mL | 28
  Day 3 ≥350 ng/mL and Day 8 <700 ng/mL | 7
  Day 3 ≥350 ng/mL and Day 8 ≥700 ng/mL | 14
  Total Day 3 ≥350 ng/mL | 21

5. Primary Outcome: Participants With a Mean POS Plasma Concentration ≥/<250 ng/mL on Day 8 and ≥/<500 ng/mL on Day 15
Description: Individual mean concentrations calculated as the average of observed concentrations at 0 hour (before the morning dose) and 5 hours after the morning dose.
Time Frame: Predose (0 hour) and 5 hours postdose on Days 8 and 15
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | POS 200 mg TID Days 1-8 Followed by POS 200 mg TID Days 9-15 | POS 200 mg TID Days 1-8 Followed by POS 400 mg BID Days 9-15 | POS 200 mg TID Days 1-8 Followed by POS 400 mg TID Days 9-15
Number analyzed (Participants) | 19 | 14 | 16
Participants
  Day 8 <250 ng/mL and Day 15 <500 ng/mL | 3 | 3 | 3
  Day 8 <250 ng/mL and Day 15 ≥500 ng/mL | 2 | 0 | 1
  Total Day 8 <250 ng/mL | 5 | 3 | 4
  Day 8 ≥250 ng/mL and Day 15 <500 ng/mL | 6 | 0 | 3
  Day 8 ≥250 ng/mL and Day 15 ≥500 ng/mL | 8 | 11 | 9
  Total Day 8 ≥250 ng/mL | 14 | 11 | 12

6. Primary Outcome: Participants With a Mean POS Plasma Concentration ≥/<350 ng/mL on Day 8 and ≥/<700 ng/mL on Day 15
Description: as for outcome 1
Time Frame: Predose (0 hour) and 5 hours postdose on Days 8 and 15
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | POS 200 mg TID Days 1-8 Followed by POS 200 mg TID Days 9-15 | POS 200 mg TID Days 1-8 Followed by POS 400 mg BID Days 9-15 | POS 200 mg TID Days 1-8 Followed by POS 400 mg TID Days 9-15
Number analyzed (Participants) | 19 | 14 | 16
Participants
  Day 8 <350 ng/mL and Day 15 <700 ng/mL | 5 | 3 | 5
  Day 8 <350 ng/mL and Day 15 ≥700 ng/mL | 1 | 0 | 2
  Total Day 8 <350 ng/mL | 6 | 3 | 7
  Day 8 ≥350 ng/mL and Day 15 <700 ng/mL | 6 | 2 | 3
  Day 8 ≥350 ng/mL and Day 15 ≥700 ng/mL | 7 | 9 | 6
  Total Day 8 ≥350 ng/mL | 13 | 11 | 9

ADVERSE EVENTS:
Groups:
- POS 200 mg TID on Days 1-8: POS 200 mg TID on Days 1-8, administered with food or oral nutritional supplements.
- POS 200 mg TID on Days 9-15: POS 200 mg TID on Days 9-15, administered with food or oral nutritional supplements.
- POS 400 mg BID on Days 9-15: POS 400 mg on Days 9-15, administered with food or oral nutritional supplements.
- POS 400 mg TID on Days 9-15: POS 400 mg TID on Days 9-15, administered with food or oral nutritional supplements.
Arm/Group | POS 200 mg TID on Days 1-8 | POS 200 mg TID on Days 9-15 | POS 400 mg BID on Days 9-15 | POS 400 mg TID on Days 9-15
Serious Adverse Events (participants affected / at risk) | 16/75 | 3/21 | 4/20 | 5/20
Other Adverse Events (participants affected / at risk) | 73/75 | 20/21 | 20/20 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POS 200 mg TID on Days 1-8 (N=75) | POS 200 mg TID on Days 9-15 (N=21) | POS 400 mg BID on Days 9-15 (N=20) | POS 400 mg TID on Days 9-15 (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute graft versus host disease in liver (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cranial neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POS 200 mg TID on Days 1-8 (N=75) | POS 200 mg TID on Days 9-15 (N=21) | POS 400 mg BID on Days 9-15 (N=20) | POS 400 mg TID on Days 9-15 (N=20)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (17) | 5 (5) | 5 (6) | 4 (4)
Tachycardia (Cardiac disorders) | 4 (5) | 0 (0) | 3 (4) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 7 (9) | 3 (4) | 1 (1) | 3 (4)
Abdominal discomfort (Gastrointestinal disorders) | 4 (6) | 0 (0) | 2 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 12 (16) | 4 (7) | 4 (5) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 15 (16) | 4 (4) | 6 (6) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 39 (83) | 10 (27) | 9 (20) | 13 (23)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 8 (11) | 4 (6) | 2 (3) | 2 (2)
Flatulence (Gastrointestinal disorders) | 11 (15) | 2 (4) | 5 (7) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 9 (12) | 4 (4) | 4 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 39 (67) | 11 (17) | 10 (14) | 12 (27)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 14 (18) | 3 (3) | 3 (3) | 5 (9)
Vomiting (Gastrointestinal disorders) | 22 (29) | 6 (10) | 5 (5) | 7 (9)
Catheter site erythema (General disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Chest pain (General disorders) | 5 (5) | 0 (0) | 2 (2) | 2 (2)
Chills (General disorders) | 14 (15) | 3 (4) | 3 (3) | 8 (8)
Mucosal inflammation (General disorders) | 20 (30) | 7 (9) | 5 (6) | 4 (10)
Oedema peripheral (General disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 33 (40) | 10 (13) | 11 (13) | 10 (12)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (17) | 0 (0) | 1 (3) | 2 (12)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Clostridial infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 4 (5) | 2 (3) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 11 (11) | 4 (4) | 4 (4) | 3 (3)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Transaminases increased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 12 (14) | 1 (1) | 4 (6) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (24) | 3 (4) | 5 (6) | 10 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 9 (9) | 3 (3) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 4 (7) | 0 (0) | 2 (3) | 2 (4)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 4 (5) | 0 (0) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 1 (1) | 3 (3) | 1 (1)
Sleep disorder (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 3 (3) | 2 (2) | 1 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 1 (1) | 3 (3) | 2 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 2 (3) | 2 (2) | 5 (6)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3) | 3 (3) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 15 (15) | 5 (5) | 6 (6) | 3 (3)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 9 (12) | 0 (0) | 4 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor and investigator will publish/present study results together with other study sites, unless written permission is obtained. The investigator provides to the sponsor 45 days prior to submission for publication/presentation, copies of abstracts or manuscripts reporting any study results. The sponsor has the right to review/comment on the data analysis and presentation regarding proprietary information, accuracy and fair blance of the information, and compliance with FDA regulations.